CLINICAL TRIAL: NCT02150278
Title: Effectiveness of an Intervention to Reduce Driving Under the Influence of Alcohol Among Drivers
Acronym: PREVENCON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Societat Catalana de Medicina Familiar i Comunitària (CAMFIC) (Unknown); Associació Catalana d'Infermeria (ACI) (Unknown); Associació Catalana d'Infermeria Familiar i Comunitària (AIFIC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PREVENCON
Record Dates: First submitted 2014-05-06; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Alcohol Consumption; Traffic Accident; Risk Perception of Driving After Alcohol Consumption
Keywords: Driving; Alcohol consumption; Risk perception
MeSH Terms: conditions — Alcohol Drinking | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brief intervention (Experimental): The brief intervention consist of one face to face minimal advice to reduce drinking-driving behavior and it was personalized according to the state of change of the patient (based on the Prochaska and DiClemente model). An additional informative pamphlet is offered to the participant. The intervention was done by the general practitioner or nurse that regularly attends the patient.
  Interventions: Behavioral: Brief intervention

INTERVENTIONS:
Behavioral: Brief intervention — The brief intervention consist of one face to face minimal advice to reduce drinking-driving behavior and it was personalized according to the state of change of the patient (based on the Prochaska and DiClemente model). An additional informative pamphlet is offered to the participant. The intervention was done by the general practitioner or nurse that regularly attends the patient.

SUMMARY:
Objectives: The main objective of this pilot study is to assess the feasibility and effectiveness of a brief intervention to reduce drinking-driving behavior.

Methods:

Design: Pilot multicentre before/after intervention study without control group. Participants: We aim to recruit, from 01/01/2013 to 01/05/2013, 212 drivers aged 18 to 65 who declared to have consumed alcohol previous to driving, at least once in the past 30 days. Intervention: Brief behavioral intervention to reduce alcohol consumption before driving. Outcomes: Frequency of driving under the influence of alcohol in the past 30 days, regular alcohol consumption (Audit-C test), level of self-efficacy and stage of change according to the Prochaska and DiClemente's Transtheoretical Model of Change, sociodemographic variables, driver's profile, chronic pathologies, long -term medications, level of self risk perception. Information will be checked against medical record. Information on a) frequency of driving under the influence of alcohol in the past 30 days, b) regular alcohol and c) level of self-efficacy and stet of change according Prochaska State will be gathered at one month and 12 month post intervention. Descriptive bivariate analysis to assess the distribution of risk elements associated to drinking-driving behavior.

Potential impact expected: This pilot project will determine the feasibility of making a brief advice intervention in drivers under the influence of alcohol in primary care.

DETAILED DESCRIPTION:
Background: Driving under the influence of alcohol is one of the main risk factors for road traffic collisions since it alters driving ability and impairs human performance. Consequently, is very important to identify those drivers who drive under the influence of alcohol; furthermore, interventions are necessary to diminish drinking-driving behavior.

Objectives: The main objective of this pilot study is to assess the feasibility and effectiveness of a brief intervention to reduce drinking-driving behavior.

Secondary objectives include:

1. To assess the effect of the intervention on stage of change and level of self-efficacy, at month 1 and 12 post-intervention.
2. To assess the feasibility of this intervention by professionals and patients.
3. To assess the effectiveness of decreasing the regular alcohol consumption at month 12 post-intervention.

Methods:

Design: Pilot multicentre before/after intervention study without control group.

Participants: We aim to recruit 212 participants. We included by random consecutive sampling drivers (with a valid driver's license) aged 18 to 65 with an open medical history in any of the 20 Primary Health Care participating centers and who declared to have consumed alcohol previous to driving, at least once in the past 30 days. Recruitment took place from xxx 2013 to xxx 213.

Intervention: Brief behavioral intervention to reduce alcohol consumption before driving.

Measurements:

At baseline, the following information will be gathered using a structured questionnaire in the face to face interview between the patient and the health professional:

1. Frequency of driving under the influence of alcohol in the past 30 days. gathered as a) the number of times that the patient drinks any amount of alcohol previous to driving and b) the amount alcohol consumed previous to driving
2. Regular alcohol consumption (Audit-C test) in units of standard drinks weekly consumed (UBE).
3. Level of self-efficacy and stage of change according to the Prochaska and DiClemente's Transtheoretical Model of Change.
4. Sociodemographic variables: age, sex, social class, educational level, marital status.
5. Driver profile: Type of driver's license, driving experience, , weekly driving time, safety behaviours, collisions (with and without injury) suffered in the past year.
6. Chronic pathologies and chronic consumption of medications associated to road traffic injuries
7. Level of self risk perception. When possible, all the information will be checked with that specified in the electronical medical record of the patient.

In order to assess the feasibility of the intervention we will undertake a survey among health professionals.

Information on a) frequency of driving under the influence of alcohol in the past 30 days, b) regular alcohol and c) level of self-efficacy and stet of change according Prochaska State will be gathered at one month and 12 month post intervention.

Analysis: A descriptive analysis of population will be performed. The distribution of risk elements associated to drinking-driving behavior will be described through bivariate analyses.

Potential impact expected:

This pilot project will determine the feasibility of making a brief advice intervention in drinking-driving behavior drivers attended in primary care.

ELIGIBILITY:
Inclusion Criteria:

* drivers with driving license of any vehicle with current validity
* People aged 18 to 65 years
* People attended Primary Health Care reported having consumed any alcohol at least one time before driving the 30 days prior

Exclusion criteria:

* People advise against that approach: severe psychiatric illnesses and terminals
* Patients with a diagnosis of alcohol dependence
* Difficulty communication language
* Unstable demographic status: People residing outside the study area, traffic situation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of driving under the influence of alcohol in the past 30 days | up to month 12 post-intervention
  We will gather a) the number of times that the patient drinks any amount of alcohol previous to driving and b) the amount alcohol consumed previous to driving

SECONDARY OUTCOMES:
Stage of change | Information will be gathered at baseline, at month 1 post-intervention, and at month 12 post-intervention.
  : Stage of change according to the Prochaska and DiClemente's Transtheoretical Model of Change, also called The Transtheoretical Model (TTM) wich assumes that individuals change habitual behaviors through a cyclical process. It includes the following stages: precontemplation, contemplation, preparation and action, among others
Regular alcohol consumption | Information will be gathered at baseline, at month 1 post-intervention, and at month 12 post-intervention.
  Regular alcohol consumption according to the Audit-C test in units of standard drinks weekly consumed (UBE). Information will be checked against patient's medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Martín_Cantera, MD, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Carlos Martin, Barcelona, Barcelona, Spain